CLINICAL TRIAL: NCT06117709
Title: Integrated Smartphone Technology to Alleviate Malignant Pain (I-STAMP): Development, Usability, and Acceptability Testing
Brief Title: Integrated Smartphone Technology to Alleviate Malignant Pain (I-STAMP) Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Andrea Enzinger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-187
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer; Pain
Keywords: Advanced Cancer; Pain management; Opioid pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — STAMP-I protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- I-STAMP Testing (Experimental): Study procedures will be conducted as follows:
  Activities 1-3: Data Collection for application development
  Activity 4: To be added with future amendment
  Interventions: Behavioral: I-STAMP

INTERVENTIONS:
Behavioral: I-STAMP — A patient-facing smartphone application that hosts participants' analgesic and laxative medications, provides pain-specific psychoeducation, collects patient reported outcomes, and provides feedback to participant symptoms.

SUMMARY:
The purpose of the study is to evaluate if the smartphone app, I-STAMP (Integrated Smartphone Technology to Alleviate Malignant Pain), helps participants with cancer pain manage symptoms and keep track of medications.

DETAILED DESCRIPTION:
The goal of this study is to develop and refine I-STAMP (Integrated Smartphone Technology to Alleviate Malignant Pain), an electronic health record-integrated mobile health (mHealth) application designed to support advanced cancer patients and care teams in pain management.

The research study procedures include screening for eligibility, surveys, and interviews. It is expected that up to 73 participants will take part in this research study. Activities 1-3 are non-interventional and will be used to collect data for application development.

Activity 4: This activity will be interventional and will be added with a future amendment.

ELIGIBILITY:
Inclusion Criteria for Participants (Activities 1a, 2a, 3a):

* Age ≥ 21 years
* Current or previous diagnosis of advanced cancer
* Current or previous experience with cancer pain

Exclusion Criteria for Participants (Activities 1a, 2a, 3a):

* Inability to understand, speak, or read English
* Any condition that would impede the patient's ability to complete study procedures such as visual impairment or significant cognitive impairment as determined by the participant's treating provider.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Usability | 2 weeks
  Patients will complete a validated 10-item system usability scale (SUS) with total scores ranging from 0-100, where a score of 100 being the best possible usability score.
E-scale Acceptability | 2 weeks
  Patients will rate overall acceptability of the application using a modified acceptability e-scale. This 6-item measure asks patients to rate the app on ease of use, understandability, enjoyment, helpfulness, time spent, and overall satisfaction, on a 1 to 5 Likert scale. Items are summed to for a total score, ranging from 6 to 30 with 30 being the highest acceptability score.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu